CLINICAL TRIAL: NCT02579304
Title: Feasibility, Safety and Diagnostic Value of Transbronchial Lung Cryobiopsy in the Work-up of Diffuse Interstitial Lung Diseases.
Brief Title: Diagnostic Value of Transbronchial Lung Cryobiopsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Yserbyt Jonas, MD, KU Leuven
Other Study IDs: UZLPNE1015
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — transbronchial lung biopsies
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: transbronchial lung cryobiopsy — bronchoscopic sampling

SUMMARY:
Evaluating the diagnostic value of transbronchial lung cryobiopsy (TBLC) as well as its procedural feasibility and safety in a prospective series of 20 patients with diffuse interstitial lung diseases (DILD) who are referred for invasive histopathological diagnostics

DETAILED DESCRIPTION:
Before one is able to state that TBLC is a technique that is an alternative for VATS biopsy, the diagnostic value of TBLC should be assessed and the value of the histopathological sampling should be compared with what is achieved by surgical lung biopsy. For this purpose direct comparison between VATS biopsy and TBLC is unavoidable. By including TBLC in the work-up of patients with DILD in which histopathological assessment is indicated (as proposed by MDD), we want to assess 3 major points of concern.

Agreement for the histopathological diagnosis between VATS biopsy and TBLC. Value of TBLC in the specific diagnosis in ILD.

ELIGIBILITY:
Inclusion Criteria:

* - Case of DILD presented at the MDD
* Referral for VATS biopsy as advised by MDD.
* Informed consent available
* Age > 18
* FVC > 50%pred
* DLCO > 40%pred
* PaO2 > 65 mmHg, pCO2 < 45 mmHg
* No exclusion criteria

Exclusion Criteria:

* - Age > 75
* PAPS >40mmHg as measured on transthoracic cardiac ultrasound
* Platelet count <100000/µl
* INR > 1.4
* BMI >30
* Diffuse bullous lung disease
* Active anti-platelet or anticoagulant treatment
* Active heart failure or unstable coronary heart disease
* Patients unfit for VATS under general anaesthesia as assessed by the surgeon and/or anesthesiologist

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: interstitial lung disease, fibrotic or non-fibrotic
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
histopathological agreement | 2 years
  Histopathological diagnostic intra-observer agreement between Video-assisted thoracosopic surgery biopsy and TBLC (kappa value)

SECONDARY OUTCOMES:
procedural safety : bleeding | periprocedural 1 hour
  incidence of bleeding (number of case)
procedural safety : bleeding (2) | periprocedural 1 hour
  severity of bleeding (grade 1-2-3)
procedural safety : bleeding (3) | periprocedural 1 hour
  duration of bleeding (seconds)
procedural safety : penumothorax | periprocedural 1 hour
  pneumothorax rate (number of cases)

CONTACTS AND LOCATIONS:
Overall Officials: jonas Yserbyt, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium